CLINICAL TRIAL: NCT05863286
Title: Assessment of Botulinum Toxin Injection for Treatment of Temporomandibular Joint Dislocation: Double-blind, Randomized, Placebo Controlled Trail Assessment of Botulinum Toxin Injection for Treatment of Temporomandibular Joint Dislocation
Brief Title: Assessment of Botulinum Toxin Injection for Treatment of Temporomandibular Joint Dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Ehab Shaaban, Amr Shaaban, BDS "Prinicipal Investigator", Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11 12 22
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Dislocation of Temporomandibular Joint TMJ; Subluxation of Temporomandibular Joint
Keywords: Botulinum Toxin; Tmj Subluxation
MeSH Terms: interventions — Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botulinum toxin type A injection in lateral pterygoid muscle (Experimental): Botulinum toxin type A vial will be reconstituted with normal saline to obtain a 10 U/0.1 ml solution, 0.25 ml of this solution containing 25 U BTX-A will be loaded in a 1-ml insulin syringe attached to a needle with 27 Gauge and 31 mm length.
  The Lateral pterygoid muscle will be approached extra orally through the space formed by the zygomatic arch and the sigmoid notch of the mandible below the center of the zygomatic arch. The needle will be advanced perpendicular to the skin with the mouth closed. The muscle is approximately 3 to 4 cm deep. Aspiration will be carried out to avoid unintentional intravascular injection. According to the assigned group, the inferior head of Lateral pterygoid muscle will be injected with BTX-A
  Interventions: Drug: Botulinum toxin type A
- Placebo "Saline 0.9%" injection in lateral pterygoid muscle (Placebo Comparator): 0.25 ml of normal saline will be loaded in a 1-ml insulin syringe attached to a needle with 27 Gauge and 31 mm length.
  The Lateral pterygoid muscle will be approached extra orally through the space formed by the zygomatic arch and the sigmoid notch of the mandible below the center of the zygomatic arch. The needle will be advanced perpendicular to the skin with the mouth closed. The muscle is approximately 3 to 4 cm deep. Aspiration will be carried out to avoid unintentional intravascular injection. According to the assigned group, the inferior head of Lateral pterygoid muscle will be injected with normal saline
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin is produced by the gram-positive, anaerobic, spore-forming bacterium Clostridium botulinum, and is one of the most lethal biological toxins known to man.
  Botulinum toxin has seven antigenically different serotypes and exerts a paralytic action by rapidly and strongly binding to presynaptic cholinergic nerve terminals. It is then internalized and ultimately inhibits the exocytosis of acetylcholine by decreasing the frequency of acetylcholine release. Without its nerve supply, the muscle fiber will deteriorate; however, the muscle will regain its strength as the nerves regenerate.
  Other Names: Botulinum Toxin

SUMMARY:
Assessment of the effect of Botulinum toxin injection on the frequency of luxation and TMJ Pain in patients with TMJ dislocation either chronic recurrent dislocation or subluxation

DETAILED DESCRIPTION:
Diagnostic procedure:

1. Patient questionnaire: a questionnaire will be recorded by the examiner including the Chief complaint, Personal data, and Medical history.
2. Consent: Informed consent will be obtained from patients to participate in the study.
3. Clinical examination: TMJ examination with specific emphasis on the TMJ regarding pain, clicking, maximum inter-incisal mouth opening, lateral excursions, and muscle examination is done (Inspection and palpation).

   o operative procedures:

   • The surgical field will be scrubbed and prepared in a standard sterile fashion using alcohol and topical anesthesia is applied at point of needle insertion

   A-Botulinum Toxin Type A injection:

   BTX-A vial will be reconstituted with normal saline to obtain a 10 U/0.1 ml solution, 0.25 ml of this solution containing 25 U BTX-A will be loaded in a 1-ml insulin syringe attached to a needle with 27 Gauge and 31 mm length.

   B-The placebo comparator Injection:

   Patients in the placebo arm will receive equivalent volumes of placebo solution (Normal Saline).

   • Procedure

   - With the patient sitting in an upright position on the dental chair, the lateral ptreygoid muscle will be approached extra orally through the space formed by the zygomatic arch and the sigmoid notch of the mandible below the center of the zygomatic arch. The needle will be advanced perpendicular to the skin with the mouth closed. The muscle is approximately 3 to 4 cm deep. Aspiration will be carried out to avoid unintentional intravascular injection.

   According to the assigned group, the inferior head of Lateral pterygoid muscle will be injected with BTX-A or normal saline

   - The patient will be instructed to remain in an upright position for 6 h (to reduce diffusion into pharyngeal muscles which may cause dysphagia and nasal regurgitation).

   - Patients will be recalled weekly during the first month, then monthly after 3 months
   * Post-operative care:

   Paracetamol 1000 mg will be prescribed as needed Any excessive mouth opening should be avoided Soft diets are advised in the first 48 hours after injection

ELIGIBILITY:
Inclusion Criteria:

1. patients with TMJ habitual or recurrent dislocation
2. Age ≥ 18 years
3. The willingness of the patient to receive relative painful injections and to follow instructions

Exclusion Criteria:

1. Patients with neurogenic cause of TMJ Hypermobility.
2. Drug-induced TMJ Hypermobility

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of luxation | 6 months
  Postoperative frequency of luxation is measured by number of luxation per day in organized sheet
Maximum Mouth opening | 6 months
  Postoperative Maximum Mouth opening is measured by digital caliper in follow up intervals" 1 week, 1 month, 3 month, 6 month"

SECONDARY OUTCOMES:
Lateral mandibular movement | 6 months
  Postoperative lateral mandibular movement " side to side movement" is measured by digital caliper in follow up intervals " 1 week, 1 month, 3 month, 6 month"

CONTACTS AND LOCATIONS:
Overall Officials: Hamida Refai, Doctor of dental science, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo university, Cairo, Elmanial, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Refai H, Altahhan O, Elsharkawy R. The efficacy of dextrose prolotherapy for temporomandibular joint hypermobility: a preliminary prospective, randomized, double-blind, placebo-controlled clinical trial. J Oral Maxillofac Surg. 2011 Dec;69(12):2962-70. doi: 10.1016/j.joms.2011.02.128. Epub 2011 Jul 16. PMID 21757278